CLINICAL TRIAL: NCT02073604
Title: Rôle de la SMA Dans la préparation Des Mouvements Uni et Bi-manuels: le Paradigme Des Mouvements en Miroir
Brief Title: Role of the SMA During Unimanual and Bimanual Movements Preparation: the Mirror Movements Paradigm
Acronym: MOMIC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C13-16; 2013-A00616-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-01-16; First posted 2014-02-27 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2016-08

CONDITIONS: Congenital Mirror Movements
Keywords: Congenital mirror movements; SMA; Movement preparation; Movement lateralization; MRI; Transcranial magnetic stimulation
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Other: Healthy volunteers
- Congenital mirror movements (Other): Patients presenting with congenital mirror movements
  Interventions: Other: Congenital mirror movements

INTERVENTIONS:
Other: Healthy volunteers — Morphological and functional brain MRI; transcranial magnetic stimulation
  Arms: Healthy volunteers
Other: Congenital mirror movements — Morphological and functional brain MRI; transcranial magnetic stimulation
  Arms: Congenital mirror movements

SUMMARY:
The aim of the project is to study the role of secondary motor area (more precisely the supplementary motor area, or SMA) during unimanual and bimanual voluntary movements externally (cue) or internally (subject's choice) triggered. In that view, we will study 3 experimental groups :

* a group of healthy volunteers (control group)
* the same group of healthy volunteers after a transient inactivation of the SMA (by the aim of repetitive trans cranial magnetic stimulation or TMS)
* a group of patients suffering from congenital mirror movements who are suspected to present a dysfunction of the SMA (according to our previous results) In each of these groups, by the aim of a serial reaction time task, we will study the influence of a SMA stimulation on the excitability of the primary motor cortex (M1) during the preparation of a voluntary movement (unimanual or bimanual). This will allow us to assess the communication between the SMA and M1 during movement preparation. Using the same task in functional imagery, we will study the activation's pattern of primary and secondary motor areas during movement preparation. This multimodal approach should allow us to better understand the synergistic functioning of these different structures involved in movement preparation. An other interesting aspect will be to determine the role of these structures in movement lateralization. Eventually, our results might allow us to precise to role of the motor preparation's dysfunction in the genesis of congenital mirror movements.

In the first place, this study aims at a better understanding of the cerebral physiology of movement preparation (which is not well known) using the mirror movements paradigm as a dysfunction model (according to our previous results). According to our hypothesis, there is a strong link between the SMA and M1 during movement preparation. This hypothesis will be assessed by the use of the same experimental task with combined neurophysiological and neuroimaging approaches, thus increasing the validity of the results obtained.

A secondary aim of this protocol is to precise the role of motor planning dysfunction in patients with congenital mirror movements. A better understanding of the mechanisms responsible for this condition is necessary in a medium-term therapeutic prospect.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 15 years and 3 months to 82 years
* Patients with congenital mirror movements without additional manifestation or malformation
* No contraindications for MRI or TMS study

Exclusion Criteria:

* Inability to provide an informed consent
* Simultaneous participation in another clinical trial
* Treatment that modulate cortical excitability (for the TMS part of the study only)

Ages: 15 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
SMA activation level and connectivity during preparation of unimanual/bimanual movements | up to 3 years

SECONDARY OUTCOMES:
SMA activation level and connectivity during preparation of unimanual/bimanual movements in congenital mirror movements patients | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ROZE, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Fédération des Maladies du Système Nerveux, Hôpital Pitié Salpétrière Paris, France 75013, Paris, France

REFERENCES:
- [Background] Chole RA. Meatoplasty using inferiorly based island pedicle flap for congenital aural atresia. Laryngoscope. 1983 Jul;93(7):954-5. doi: 10.1288/00005537-198307000-00025. No abstract available. PMID 6865634